CLINICAL TRIAL: NCT03045653
Title: Efficacy and Safety of High Dose Tamoxifen to Advanced Hormone Receptor-High Expressed Endocrine Therapy Resisted Breast Cancer
Brief Title: Efficacy of High Dose Tamoxifen to Advanced Hormone Receptor-High Expressed Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, professer, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-009
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer Metastatic
Keywords: Breast Cancer; high dose Tamoxifen; endocrine therapy; Hormone Receptor Positive Malignant Neoplasm of Breast; Tamoxifen; Breast Cancer Metastatic
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): receiving a treatment of tamoxifen 100 mg/d or high-dose Tamoxifen(100 mg/d ) plus chemotherapy
  Interventions: Drug: Tamoxifen Oral Product

INTERVENTIONS:
Drug: Tamoxifen Oral Product — Tamoxifen 100 mg/d or high-dose Tamoxifen(100 mg/d ) plus chemotherapy

SUMMARY:
Background: Endocrine therapy is an effective and safe treatment for hormone receptor positive breast cancer. Unfortunately , endocrine treatment resistance occurs and there is an urgent need for treatment alternative. Laboratory researches and clinical case reports indicate that hormone receptor-high expressed breast cancer patients may potentially benefit from high-dose Tamoxifen or high-dose Tamoxifen plus chemotherapy , providing a new option for treatment strategy.

Aim: To explore the efficacy and safety of high-dose Tamoxifen to standard hormone receptor-high expressed endocrine therapy resisted breast cancer.

Methods: Eligible patients will be treated with tamoxifen 100 mg/d or high-dose Tamoxifen(100 mg/d ) plus chemotherapy. Blood and tumor samples will be obtained from the patients.Evaluate curative effect every 3 months.

Primary endpoint: progression-free survival (PFS). Secondary endpoints: objective response rate (ORR), clinical benefit rate (CBR), overall survival (OS) and safety.

Exploratory endpointsincluded the efficacy predictive value of the 18F-FES SUVmax.

ELIGIBILITY:
Inclusion Criteria:

- Female ≥ 18 years, ≤70 years. ECOG 0-1 with no deterioration over previous 2 weeks Minimum life expectancy 3 months Histological confirmation of hormone receptor-high expressed breast cancer(IHC:ER ≥60% and PR≥60%) on primary tumour at diagnosis/on biopsy of metastasis Histological confirmation of HER2 negative breast cancer on primary tumour at diagnosis/on biopsy of a metastasis The disease-free time of relapsed patients is more than 12 months Once received standard hormone treatment and progressed Clinical or histological confirmation of metastatic or locally advanced disease not amenable to curative surgical resection At least one evaluative focus according to RECIST creterion or non-measurable disease but only bone metastasis Adequate bone marrow and organ function Progressive disease whilst receiving endocrine therapy for locally advanced or metastatic BC or relapsed with metastatic disease whilst receiving endocrine therapy Radiological or objective clinical evidence of recurrence or progression on or after last systemic therapy prior to enrolment

* 4 prior lines of endocrine therapy for ABC
* 3 line of cytotoxic chemotherapy for ABC Suitable for further endocrine therapy Availability of archival tumour sample or fresh biopsy Informed consent Normal organ function

Exclusion Criteria:

* Last dose chemotherapy, immunotherapy targeted therapy, biological therapy or tumour embolisation <21 days prior to study treatment Last dose of palliative radiotherapy <7 days prior to study treatment Rapidly progressive visceral disease not suitable for further endocrine therapy Spinal cord compression or brain/meningeal metastases unless asymptomatic, treated and stable and not requiring steroids for ≥ 4 weeks study treatment Creatinine clearance <30 ml/min. Patients with creatinine clearance <50 mL/min will start at a permanently reduced vandetanib dose of 200 mg.

Major surgery (excluding placement of vascular access) within 4 weeks before study treatment Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and HIV With the exception of alopecia, any unresolved toxicities from previous therapy greater than CTCAE grade 1 before study treatment Elevated ALP in absence of bone metastasis Evidence of dementia, altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent Participation in another study with investigational product during last 30 days Inability or unwillingness to comply with study procedures, including inability to take regular oral medication

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyu Yuan, Principal Investigator — Sun-yatsen University Cancer center
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: receiving a treatment of tamoxifen 100 mg/d
Period: Overall Study
Arm/Group | Treatment Arm
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 45 [27 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Time Frame: 36months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 30
months | 5 [2.6 to 7.3]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 7/30
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=30)
fatigue (General disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03045653/Prot_SAP_000.pdf